CLINICAL TRIAL: NCT01670955
Title: A Prospective Phase II/III Randomized, Blinded Study to Demonstrate the Safety and Effectiveness of Jobelyn ( a Herbal Preparation ) in Pre-operative Management of Anaemia in Gynaecological Patients
Brief Title: The Safety and Effectiveness of Jobelyn in Pre-operative Management of Anaemia in Gynaecological Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lagos State University (Other)
Collaborators: Health Forever Product Limited. Lagos, Nigeria (Unknown)
Responsible Party: Principal Investigator, Dr. A. Tayo, CONSULTANT IN THE DEPARTMENT OF GYNAECOLOGY AND OBSTETRICS, LASUTH, Lagos State University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: LASUTH/08/2012
Record Dates: First submitted 2012-08-18; First posted 2012-08-23 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Anemia
Keywords: Anemia; preoperative; gynecological patients; Sorghum bicolor; Packed Cells Volume
MeSH Terms: conditions — Anemia | interventions — ferrous sulfate; Folic Acid; Iron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Jobelyn + Ferrous Sulphate + Folic Acid (Active Comparator): Caps Jobelyn 250mg, 12 hourly + Ferrous Sulphate 600mg thrice daily + Folic Acid 5mg daily
  Interventions: Dietary Supplement: Jobelyn; Drug: Ferrous Sulphate + Folic Acid
- Ferrous Sulphate + Folic Acid (Active Comparator): Ferrous Sulphate 600mg, thrice daily + Folic Acid, 5mg daily
  Interventions: Drug: Ferrous Sulphate + Folic Acid

INTERVENTIONS:
Dietary Supplement: Jobelyn — Jobelyn is a sorghum bicolor extract marketed as dietary supplement
  Other Names: Sorghum bicolor extract
  Arms: Jobelyn + Ferrous Sulphate + Folic Acid
Drug: Ferrous Sulphate + Folic Acid — Ferrous Sulphate 600mg, thrice daily + Folic Acid, 5mg daily
  Other Names: Iron Tablets

SUMMARY:
PROTOCOL FOR THE STUDY OF THE SAFETY AND EFFICACY OF JOBELYN, IN THE PREOPERATIVE MANAGEMENT OF ANAEMIA IN GYNAECOLOGICAL PATIENTS

DETAILED DESCRIPTION:
It has long been known that anaemia increases the risk of death and complications in patients who have cardiovascular surgery, but results of a recent study show that these risks are increased in patients with anaemia who undergo various types of surgery, including gynaecological procedures.

Compared with patients without anaemia, the risk of death within 30 days after surgery was 42% higher among patients with anaemia. In addition, patients with anemia were 35% more likely to experience cardiac, respiratory, urinary, and wound complications as well as sepsis and blood clots.

Because even mild anaemia increases the risk of postoperative morbidity in patients undergoing major non-cardiac surgery, doctors need to consider preoperative treatment of anaemia when possible. More research is needed to establish the efficacy, safety and cost-effectiveness of pre-operative anaemia management.

One of the major clinical issues in many gynaecological patients in Nigeria is that of optimizing the packed cell volume before surgery. Anaemia could be traced to multiple factors notable of which are high prevalence of infection, worm infestation and malnutrition (R). In other to reduce the waiting time and reduce morbidity and mortality associated with surgery, it is important to correct the packed cell volume adequately before surgery.

The traditional method of correcting PCV involves the use of 'routine' haematinics such as Ferrous sulphate, Folic acid and Multivitamin. This is in addition to dietary advice. While the efficacy of these drugs has been well acknowledged in clinical practice, there is dearth of literatures on their specific influence on haematological parameters. Majority of Nigerians are gradually having a change of perception about traditional medicines with gradual shift towards their use. It is believed that traditional drugs act faster and more effective than other orthodox drugs in conventional use. One of such area is in the correction of anaemia.

Sorghum bicolor, a grain long used in Africa for its high nutritional value also exhibits strong antioxidant properties and antiinflammatory effects. The traditional preparation of Sorghum bicolor has an oxygen radical absorbance capacity (ORAC) OF 37,622 micro mole TE/g. This is much higher than other botanical preparations. Complementing the antioxidant properties, Sorghum bicolor also exhibits anti inflammatory effects and demonstrated selective COX-2 inhibition, providing effective reduction in inflammation without residual side effects.

Sorghum bicolor extract has been shown to increase the haematocrit and haemoglobin level and reduce the white cell count in trypanosome brucei brucei induced anaemia in experimental rabbits. These effects were conclusive within 49 days of experimentation. Animals sacrificed after the administration of lethal dose Jobelyn were shown to have congestion of the liver, kidneys and lungs. This might be as a result of direct effect on these organs or a sign of cardiotoxicity. However there is a wide therapeutic range.

Sorghum bicolor is the proprietary name for the product intended to treat sickle cell disease. It is exactly the same as jobelyn which is currently marketed as a nutritional supplement. Jobelyn is marketed in 250mg capsules of sorghum bicolor leaf extract. The product is widely marketed in the United States and in Nigeria. Many pregnant women have been using it regularly for a long time without any report of adverse effect.

The sorghum bicolor extract is expected to increase the haematocrit of' pregnant women within a short time.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate anaemia
* Asymptomatic severe anaemia
* Non life threatening gynaecological condition

Exclusion Criteria:

* Failure to give informed consent
* Symptomatic severe anaemia
* Pregnancy
* Malignancies and Chronic inflammatory disease

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Anaemia | 3 months
  Change in haematological parameters

SECONDARY OUTCOMES:
morbidity | 3 months
  Reduced postoperative morbidity

OTHER OUTCOMES:
Hospital Stay | 3 months
  Duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Adetokunbo O Tayo, M.D., Principal Investigator — Lagos State University
Locations (1):
- Lagos State University Teaching Hospital, Ikeja, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brohan M, Jerkovic V, Collin S. Potentiality of red sorghum for producing stilbenoid-enriched beers with high antioxidant activity. J Agric Food Chem. 2011 Apr 27;59(8):4088-94. doi: 10.1021/jf1047755. Epub 2011 Mar 7. PMID 21381750
- [Background] Geera B, Ojwang LO, Awika JM. New highly stable dimeric 3-deoxyanthocyanidin pigments from sorghum bicolor leaf sheath. J Food Sci. 2012 May;77(5):C566-72. doi: 10.1111/j.1750-3841.2012.02668.x. Epub 2012 Apr 10. PMID 22489620
- [Background] Kayode AP, Nout MJ, Linnemann AR, Hounhouigan JD, Berghofer E, Siebenhandl-Ehn S. Uncommonly high levels of 3-deoxyanthocyanidins and antioxidant capacity in the leaf sheaths of dye sorghum. J Agric Food Chem. 2011 Feb 23;59(4):1178-84. doi: 10.1021/jf103963t. Epub 2011 Jan 25. PMID 21322653
- [Background] Yang L, Browning JD, Awika JM. Sorghum 3-deoxyanthocyanins possess strong phase II enzyme inducer activity and cancer cell growth inhibition properties. J Agric Food Chem. 2009 Mar 11;57(5):1797-804. doi: 10.1021/jf8035066. PMID 19256554
- [Background] Shih CH, Siu SO, Ng R, Wong E, Chiu LC, Chu IK, Lo C. Quantitative analysis of anticancer 3-deoxyanthocyanidins in infected sorghum seedlings. J Agric Food Chem. 2007 Jan 24;55(2):254-9. doi: 10.1021/jf062516t. PMID 17227050
- [Background] Camargo Filho I, Cortez DA, Ueda-Nakamura T, Nakamura CV, Dias Filho BP. Antiviral activity and mode of action of a peptide isolated from Sorghum bicolor. Phytomedicine. 2008 Mar;15(3):202-8. doi: 10.1016/j.phymed.2007.07.059. Epub 2007 Sep 24. PMID 17890069
- [Background] Burdette A, Garner PL, Mayer EP, Hargrove JL, Hartle DK, Greenspan P. Anti-inflammatory activity of select sorghum (Sorghum bicolor) brans. J Med Food. 2010 Aug;13(4):879-87. doi: 10.1089/jmf.2009.0147. PMID 20673059
- [Background] Park JH, Darvin P, Lim EJ, Joung YH, Hong DY, Park EU, Park SH, Choi SK, Moon ES, Cho BW, Park KD, Lee HK, Kim MJ, Park DS, Chung IM, Yang YM. Hwanggeumchal sorghum induces cell cycle arrest, and suppresses tumor growth and metastasis through Jak2/STAT pathways in breast cancer xenografts. PLoS One. 2012;7(7):e40531. doi: 10.1371/journal.pone.0040531. Epub 2012 Jul 6. PMID 22792362
- [Background] Wu L, Huang Z, Qin P, Yao Y, Meng X, Zou J, Zhu K, Ren G. Chemical characterization of a procyanidin-rich extract from sorghum bran and its effect on oxidative stress and tumor inhibition in vivo. J Agric Food Chem. 2011 Aug 24;59(16):8609-15. doi: 10.1021/jf2015528. Epub 2011 Jul 29. PMID 21780844
- [Background] Devi PS, Kumar MS, Das SM. Evaluation of antiproliferative activity of red sorghum bran anthocyanin on a human breast cancer cell line (mcf-7). Int J Breast Cancer. 2011;2011:891481. doi: 10.4061/2011/891481. Epub 2011 Oct 16. PMID 22312562
- [Background] Awika JM, McDonough CM, Rooney LW. Decorticating sorghum to concentrate healthy phytochemicals. J Agric Food Chem. 2005 Aug 10;53(16):6230-4. doi: 10.1021/jf0510384. PMID 16076098